CLINICAL TRIAL: NCT00814840
Title: Triple-Site Versus Standard Cardiac Resynchronization Therapy (TRUST CRT) Randomized Trial
Brief Title: Efficiency Study of Triple-Site Cardiac Resynchronization in Patients With Heart Failure
Acronym: TRUST CRT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Radoslaw Lenarczyk, Primary Investigator, Silesian Centre for Heart Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SilesianCHD-KNW-6501-3/08
Record Dates: First submitted 2008-12-22; First posted 2008-12-25 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Congestive Heart Failure; Heart Disease
Keywords: Heart failure; Dyssynchrony; Cardiac resynchronization; Triple-site pacing
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple-site group (Active Comparator): Triple-site resynchronization group
  Interventions: Device: Triple-site cardiac resynchronization
- Standard resynchronization group (Active Comparator): Standard (double-site) resynchronization group
  Interventions: Device: Cardiac resynchronization pacemaker (InSync Sentry or Concerto, Medtronic, Minneapolis, MN,USA) with two intracardiac leads

INTERVENTIONS:
Device: Cardiac resynchronization pacemaker (InSync Sentry or Concerto, Medtronic, Minneapolis, MN,USA) with two intracardiac leads — Cardiac resynchronization with two intraventricular leads: one in the right ventricle and one in the left ventricle (via the coronary sinus)
  Arms: Standard resynchronization group
Device: Triple-site cardiac resynchronization — Cardiac resynchronization pacemaker (InSync Sentry or Concerto, Medtronic, Minneapolis, MN,USA) with three intraventricular leads: one in the right ventricle and two in the left ventricle (via the coronary sinus). Two left ventricular leads connected with Y-connector (Lead Adaptor 2827, Medtronic, Minneapolis, MN, USA)
  Arms: Triple-site group

SUMMARY:
The purpose of this study is to assess the efficiency of permanent biventricular pacing using three ventricular leads in terms of reduction in adverse cardiac events rates, improvement in cardiac capacity and patients' functional status in subjects with congestive heart failure and a physiologic (sinus) rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more,
* Congestive heart failure (HF) in NYHA class III-IV within last 90 days despite optimal medical treatment,
* Left ventricular ejection fraction (EF) <=35% measured with echocardiography,
* Sinus rhythm >90% of the time in 24-h Holter monitoring 1-3 days prior to randomization,
* Inter- or intraventricular mechanical dyssynchrony ≥40ms measured with pulse Doppler and tissue Doppler echocardiography,
* Optimal pharmacotherapy during the last 90 days,
* Signed informed, written consent.

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Unstable HF requiring hospitalization with intravenous inotropic drugs within last 90 days,
* Myocardial infarction, percutaneous/surgical revascularization or any cardiosurgical procedure within 90 days prior to randomization,
* Stroke within last 90 days,
* History of chronic or persistent atrial fibrillation, flutter, tachycardia,
* Acute myocarditis,
* Implanted previously pacemaker, ICD or CRT-device,
* Participation in a concurrent trial that could confuse the results of this study,
* Mechanical right heart valve,
* Prior heart transplant,
* Valvular disease that is indication for valve surgery,
* Coronary heart disease if percutaneous or surgical revascularization is indicated and possible,
* Any state, apart from HF, that limits the estimated survival time to <1 year,
* Unwillingness or inability to understand the nature of the study, to participate or to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Combined end-point of alive status, freedom from hospitalization for HF or heart transplantation, relative ≥10% increase in LV ejection fraction, ≥10% in VO2max and ≥10% in 6MWD. | six months

SECONDARY OUTCOMES:
The occurrence of major adverse cardiovascular events (hospitalization for exacerbated HF requiring modification of pharmacotherapy, heart transplant or death). | five years

CONTACTS AND LOCATIONS:
Overall Officials: Radosław Lenarczyk, M.D., Principal Investigator — First Department of Cardiology, Silesian Medical University, Silesian Center for Heart Diseases; Zbigniew Kalarus, M.D., Study Chair — First Department of Cardiology, Silesian Medical University, Silesian Center for Heart Diseases
Locations (1):
- First Department of Cardiology, Silesian Medical University, Silesian Center for Heart Diseases, Zabrze, Poland

REFERENCES:
- [Background] Lenarczyk R, Kowalski O, Kukulski T, Pruszkowska-Skrzep P, Sokal A, Szulik M, Zielinska T, Kowalczyk J, Pluta S, Sredniawa B, Musialik-Lydka A, Kalarus Z. Mid-term outcomes of triple-site vs. conventional cardiac resynchronization therapy: a preliminary study. Int J Cardiol. 2009 Mar 20;133(1):87-94. doi: 10.1016/j.ijcard.2007.12.009. Epub 2008 Feb 19. PMID 18242737
- [Background] Lenarczyk R, Kowalski O, Kukulski T, Szulik M, Pruszkowska-Skrzep P, Zielinska T, Kowalczyk J, Pluta S, Duszanska A, Sredniawa B, Musialik-Lydka A, Kalarus Z. Triple-site biventricular pacing in patients undergoing cardiac resynchronization therapy: a feasibility study. Europace. 2007 Sep;9(9):762-7. doi: 10.1093/europace/eum140. Epub 2007 Jul 13. PMID 17631515
- [Background] Leclercq C, Gadler F, Kranig W, Ellery S, Gras D, Lazarus A, Clementy J, Boulogne E, Daubert JC; TRIP-HF (Triple Resynchronization In Paced Heart Failure Patients) Study Group. A randomized comparison of triple-site versus dual-site ventricular stimulation in patients with congestive heart failure. J Am Coll Cardiol. 2008 Apr 15;51(15):1455-62. doi: 10.1016/j.jacc.2007.11.074. PMID 18402900
- [Background] Lenarczyk R, Kowalski O, Sredniawa B, Pruszkowska-Skrzep P, Pluta S, Sokal A, Kukulski T, Stabryla-Deska J, Wozniak A, Kowalczyk J, Zielinska T, Mazurek M, Streb W, Zembala M, Kalarus Z. Triple-site versus standard cardiac resynchronization therapy study (TRUST CRT): clinical rationale, design, and implementation. J Cardiovasc Electrophysiol. 2009 Jun;20(6):658-62. doi: 10.1111/j.1540-8167.2008.01394.x. PMID 19635069
- [Result] Lenarczyk R, Kowalski O, Sredniawa B, Pruszkowska-Skrzep P, Mazurek M, Jedrzejczyk-Patej E, Wozniak A, Pluta S, Glowacki J, Kalarus Z. Implantation feasibility, procedure-related adverse events and lead performance during 1-year follow-up in patients undergoing triple-site cardiac resynchronization therapy: a substudy of TRUST CRT randomized trial. J Cardiovasc Electrophysiol. 2012 Nov;23(11):1228-36. doi: 10.1111/j.1540-8167.2012.02375.x. Epub 2012 May 31. PMID 22651239
- [Derived] Lenarczyk R, Jedrzejczyk-Patej E, Mazurek M, Szulik M, Kowalski O, Pruszkowska P, Sokal A, Sredniawa B, Boidol J, Kowalczyk J, Podolecki T, Mencel G, Kalarus Z. Quality of life in cardiac resynchronization recipients: association with response and impact on outcome. Pacing Clin Electrophysiol. 2015 Jan;38(1):8-17. doi: 10.1111/pace.12523. Epub 2014 Oct 15. PMID 25319879
- [Derived] Kowalczyk J, Lenarczyk R, Kowalski O, Podolecki T, Francuz P, Pruszkowska-Skrzep P, Szulik M, Mazurek M, Jedrzejczyk-Patej E, Sredniawa B, Kalarus Z; Triple-Site Versus Standard Cardiac Resynchronization Trial (TRUST CRT) Investigators. Contrast-induced acute kidney injury in patients undergoing cardiac resynchronization therapy-incidence and prognostic importance. Sub-analysis of data from randomized TRUST CRT trial. J Interv Card Electrophysiol. 2014 Jun;40(1):1-8. doi: 10.1007/s10840-014-9887-x. Epub 2014 Mar 14. PMID 24626998
- [Derived] Boidol J, Sredniawa B, Kowalski O, Szulik M, Mazurek M, Sokal A, Pruszkowska-Skrzep P, Kukulski T, Kalarus Z, Lenarczyk R; Triple-Site Versus Standard Cardiac Resynchronisation Trial (TRUST CRT) Investigators. Many response criteria are poor predictors of outcomes after cardiac resynchronization therapy: validation using data from the randomized trial. Europace. 2013 Jun;15(6):835-44. doi: 10.1093/europace/eus390. Epub 2013 Mar 13. PMID 23487543